CLINICAL TRIAL: NCT01152138
Title: COCHISE Pilot Study: Closed vs Open Cells Stent for High Risk Percutaneous Coronary Interventions in ST Elevation Acute Myocardial Infarction
Brief Title: Closed Versus Open Cells Stent for Acute Myocardial Infarction
Acronym: COCHISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alessandro Sciahbasi (Other)
Responsible Party: Sponsor-Investigator, Alessandro Sciahbasi, Medical doctor, Policlinico Casilino ASL RMB
Organization: Policlinico Casilino ASL RMB (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COCHISE
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2012-05-17 (Estimated); Status verified 2012-05

CONDITIONS: Acute Myocardial Infarction; Primary Percutaneous Coronary Intervention
Keywords: Acute myocardial infarction; Closed cell stent; Open cell stent; primary percutaneous coronary intervention
MeSH Terms: interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Cell Stent (Active Comparator): Open cell stent (Driver™ or Integrity™,Medtronic), routinely employed during percutaneous coronary interventions for ST elevation acute myocardial infarction
  Interventions: Device: Open cells stent
- Closed Cell Stent (Active Comparator): Closed cell stent (Presillion Plus™, Cordis), routinely employed during percutaneous coronary interventions for ST elevation acute myocardial infarction
  Interventions: Device: Closed Cells Stent

INTERVENTIONS:
Device: Open cells stent — Cobalt Chromium Stent with open cell design
  Other Names: Driver Stent, Medtronic; Integrity Stent, Medtronic
  Arms: Open Cell Stent
Device: Closed Cells Stent — Cobalt Chromium stent with closed cell design
  Other Names: Presillion Plus Stent, Cordis
  Arms: Closed Cell Stent

SUMMARY:
The aim of this study is to determine whether a closed cell stent design may reduce distal embolization and no reflow during primary percutaneous coronary intervention (PPCI) for acute ST-elevation acute myocardial infarction (STEMI) compared to an open cell stent design. The study population will include all consecutive patients admitted for acute STEMI and treated with PPCI within 12 hours from symptom onset.

DETAILED DESCRIPTION:
BACKGROUND Primary percutaneous coronary intervention (PPCI) represents the "gold standard" in the current management of patients with acute ST-elevation myocardial infarction (STEMI). Indeed, PPCI is associated with a rapid restore of coronary flow and with a better outcome compared to pharmacological therapy. However in a sizable proportion of patients PPCI achieves only epicardial coronary artery reperfusion but not myocardial reperfusion, a condition known as no-reflow. A series of consistent data has clearly shown that no-reflow has a strong negative impact on outcome, negating the potential benefit of PPCI. No-reflow may be caused by the variable combination of 4 pathogenetic components: 1) distal atherothrombotic embolization; 2) ischemic injury; 3) reperfusion injury; and 4) susceptibility of coronary microcirculation to injury. In particular during PPCI emboli of different sizes can originate from fissurated atherosclerotic plaques and occlude the microvascular bed. Several pharmacological, mechanical or technical strategies have been proposed for the prevention and treatment of distal embolization and coronary no-reflow with variable results, but there are no data addressing the possible effect of different stent designs on the distal embolization of thrombotic fragments.

Coronary stents can be divided in open cell or closed cell stents according to their design. Typically, the number and arrangement of bridge connectors differentiate open-cell from closed-cell designs. If adjacent ring segments are connected at every possible junction, the design is classified as closed cell. If some or all of the connecting junction points are removed, the design is classified as open cell. Such a design inherently allows for more flexion between adjacent rings, because fewer connection points allow for greater flexion and conformability. The flexion benefits of an open-cell design have a cost in scaffolding uniformity, just as the scaffolding benefits of a closed-cell design have a cost in flexion and conformability. A previous study, performed in patients who underwent carotid stenting, showed a significant reduction in distal embolization associated with the use of closed cell stents compared to open cell stents. However there are no study comparing the open or closed stent design during percutaneous coronary intervention particularly in condition at high risk of embolization as acute myocardial infarction.

STUDY HYPOTHESIS AND OBJECTIVES The aim of this study is to determine whether a closed cell stent design may reduce distal embolization and no reflow during PPCI for acute STEMI compared to an open cell stent design. The study population will include all consecutive patients admitted in our hospital for acute STEMI and treated with PPCI within 12 hours from symptom onset.

METHODS Design This study will be a prospective, randomized trial.

Patient selection Eligibility criteria: patients with an age > 18 years with acute STEMI treated with PPCI within 12 hours from symptom onset and who agree and provide written informed consent. STEMI is defined as chest pain associated with ST-elevation of 1 mm or more in two or more contiguous leads or new left bundle-branch block within 12 hours after the onset of chest pain.

Exclusion criteria will be: implanted stent with diameter < 2.5 mm, cardiogenic shock, time from pain onset to PPCI >12 hours, previous thrombolytic therapy (rescue PPCI), inability to provide informed consent.

Subjects who meet all of the inclusion criteria and none of the exclusion criteria may be enrolled into the study.

Interventional procedure All patients enrolled in this randomized study should be treated according to the standard of care of our centre and according to guidelines.

Pharmacological treatment. At admission and before the procedure all patients will be treated with 500 mg of chewable aspirin, with 600 mg of clopidogrel and with 5000 U of unfractionated heparin i.v. Additional intravenous heparin will be administered during the procedure to maintain an activated clotting time of 200-250 seconds with the use of glycoprotein IIb/IIIa inhibitors or 250-300 seconds without the administration of glycoprotein IIb/IIIa inhibitors. The administration of glycoprotein IIb/IIIa inhibitors (preferably intracoronary abciximab) will be left to the operator's discretion but is significantly encouraged. At the end of the procedure and before the final angiography a dose of 1 µg of nitrate i.c. will be administrated.

After the procedure in all cases heparin administration will be interrupted and patients will be treated with low dose of aspirin (100 mg/day) and clopidogrel (75 mg/day).

Procedure. Direct stenting is encouraged, but the use of predilation is left to operator's discretion. The use of manual thrombectomy before stenting or predilation is mandatory in case of Thrombolysis in myocardial infarction (TIMI) flow ≤1 or high thrombus burden after crossing the lesion with the wire. In all cases an effort should be made to use a single stent whenever possible. All stent will be deployed at 14 atmosphere for 30 seconds and then in all cases an angiography will be performed. Post-dilatation with over expansion of the stent is discouraged but it is allowed in cases of sub-optimal angiographic results.

Stent. Two different stent design will be employed: a closed cell stent (Presillion Plus™, Cordis) and two open cell stents (Driver™ or Integrity™, Medtronic).

Randomization. Eligible patients will be randomly assigned in a 1:1 ratio to receive either the closed cell stent or the open stent cell. Allocation to one of the two stent will be made by means of sealed envelopes containing a concealed computer-generated random sequence which was set in blocks of 20.

In-hospital assessment and clinical follow-up Laboratory tests: patients will undergo pre-procedural, 12, 24 and 48 hours blood draws to measure creatine kinase (CK), CK-myocardial band (CK-MB) mass, and troponin T as routinely scheduled for all patients in our centre.

Electrocardiogram: A 12 lead electrocardiogram (ECG) will be recorded before and after the procedure to evaluate the ST resolution

END-POINTS Primary end-point: the primary end-point will be the corrected TIMI frame count at the end of the procedure defined as the number of frames required to opacify standardized angiographic landmarks and normalized for vessel length and a composite angiographic and electrocardiographic end-point including angiographic events such as distal embolization, slow-flow (decrease in flow from TIMI 3 to TIMI 2) or no-reflow (decrease in flow from TIMI 2 or 3 to TIMI 0 or 1) and a binary ECG criterion of microvascular reperfusion injury as defined by the presence of persistent (>50% of initial value) ST-segment elevation 30 to 60 min after completion of the procedure as previously described.

Secondary end-points: Secondary end-points will be: the corrected TIMI frame count after stent deployment; a composite angiographic end-point including angiographic events such as distal embolization, slow-flow (decrease in flow from TIMI 3 to TIMI 2) or no-reflow (decrease in flow from TIMI 2 or 3 to TIMI 0 or 1) after stent deployment; the infarct size detect by myocardial enzyme release.

Tertiary end-points: in hospital major adverse cardiac events (MACE) (death, reinfarction, target lesion revascularization)

ELIGIBILITY:
Inclusion Criteria:

* patients with an age > 18 years with acute ST elevation myocardial infarction (STEMI) treated with primary percutaneous coronary intervention (PPCI) within 12 hours from symptom onset and who agree and provide written informed consent. STEMI is defined as chest pain associated with ST-elevation of 1 mm or more in two or more contiguous leads or new left bundle-branch block within 12 hours after the onset of chest pain

Exclusion Criteria:

* implanted stent with diameter < 2.5 mm
* cardiogenic shock
* time from pain onset to PPCI >12 hours
* previous thrombolytic therapy (rescue PPCI)
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Post procedural angiographic evaluation | whithin 1 day
  The corrected Thrombolysis In Myocardial Infarction (TIMI) frame count at the end of the procedure defined as the number of frames required to opacify angiographic landmarks and normalized for vessel length and a composite end-point including angiographic events such as distal embolization, slow-flow (decrease in flow from TIMI 3 to TIMI 2) or no-reflow (decrease from TIMI 2 or 3 to TIMI 0 or 1) and a binary electrocardiographic criterion of microvascular injury as defined by the presence of persistent (>50% of initial value) ST-segment elevation 30-60 min after procedure

SECONDARY OUTCOMES:
Post stent angiographic results and in hospital MACE | whithin 7 days
  The corrected Thrombolysis In Myocardial Infarction (TIMI) frame count after stent deployment; a composite angiographic end-point including angiographic events such as distal embolization, slow-flow (decrease in flow from TIMI 3 to TIMI 2) or no-reflow (decrease in flow from TIMI 2 or 3 to TIMI 0 or 1) after stent deployment; the infarct size detect by myocardial enzyme release, in hospital major adverse cardac events (MACE)(death, reinfarction, target lesion revascularization)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Sciahbasi, MD, Principal Investigator — Policilnico Casilino - ASL RMB
Locations (2):
- Italy (2):
  - UOC Cardiologia - Policlinico Casilino - ASL RMB, Rome
  - UOC Cardiologia - Ospedale Belcolle, Viterbo